CLINICAL TRIAL: NCT07287631
Title: Clinical Evaluation of Precision for the Potassium and Ionized Calcium Tests Using the i-STAT CG8+ Cartridge With the i-STAT 1 Analyzer for Capillary Specimens
Brief Title: Clinical Evaluation of Precision for the Potassium and Ionized Calcium Tests in Capillary Specimens
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Point of Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CS-2025-0002
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-08

CONDITIONS: Hematologic Tests
Keywords: Potassium (K) and ionized calcium (iCa)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Precision of potassium (K) and ionized calcium (iCa) tests in capillary blood (Other): Precision evaluation of the i-STAT K test and the i-STAT iCa test using i-STAT CG8+ cartridge on i-STAT 1 analyzer with capillary specimens from each subject enrolled in the study.
  Interventions: Diagnostic Test: Capillary blood draw

INTERVENTIONS:
Diagnostic Test: Capillary blood draw — Capillary whole blood specimens collected from fingerstick(s) will be collected from each enrolled subject with blood collection capillary tubes.

SUMMARY:
Assess precision of the i-STAT potassium (K) and ionized calcium (iCa) tests using i-STAT CG8+ cartridge on the i-STAT 1 analyzer.

DETAILED DESCRIPTION:
The objective of this study is to assess the precision of the i-STAT K and iCa tests using the IUO i-STAT CG8+ cartridge on the i-STAT 1 analyzer using results from two separate capillary specimens from each subject enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated consent form (waiver/alteration of consent, waiver of documentation of consent may be acceptable, per IRB)
2. ≥ 18 years of age

Exclusion Criteria:

1. Previous enrollment in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 425 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Precision assessment | Thirty (30) minutes from subject enrollment to the end of the blood draw and testing.
  Assess the precision of the i-STAT potassium (K) and ionized calcium (iCa) tests in mmol/L with the investigational use only (IUO) i-STAT CG8+ cartridge on the i-STAT 1 analyzer using results from capillary specimens from each subject enrolled in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Manish Gupta, MS, MBA, Study Director — Abbott Point of Care
Locations (3):
- United States (3):
  - University of New Mexico, Albuquerque, New Mexico
  - Penn State Health Milton S. Hershey Medical Center (Hershey), Hershey, Pennsylvania
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No